CLINICAL TRIAL: NCT02028975
Title: Search for Biological Markers of Orosensory Perception of Fatty Acids in Healthy Subjects and Possible Modifications in Patients With Type 2 Diabetes and in Obese Non-diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Other
Other Study IDs: VERGES 2009
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes or Obesity Without Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linoleic Acid

ARMS (3):
- Patients with type 2 diabetes (Other)
  Interventions: Other: Measure the threshold of detection for linoleic acid; Other: Oral stimulation tests; Other: Venous blood samples; Other: Samples for genetic studies (ancillary study)
- Obese patients without diabetes (Other)
  Interventions: Other: Measure the threshold of detection for linoleic acid; Other: Oral stimulation tests; Other: Venous blood samples; Other: Samples for genetic studies (ancillary study)
- Healthy volunteers (Other)
  Interventions: Other: Measure the threshold of detection for linoleic acid; Other: Oral stimulation tests; Other: Venous blood samples; Other: Samples for genetic studies (ancillary study)

INTERVENTIONS:
Other: Measure the threshold of detection for linoleic acid
Other: Oral stimulation tests
Other: Venous blood samples
Other: Samples for genetic studies (ancillary study)

SUMMARY:
Animal studies have shown that stimulation of the lingual lipid-receptor, CD 36, is accompanied by the rapid secretion of hormones in the digestive tract (incretines). We aim to determine in healthy humans whether the orosensory perception of fatty acids is followed by a modification in plasma levels of digestive tract hormones (cholecystokinin, GIP, GLP-1, secretin, pancreatic peptide, peptide YY, insulin) and metabolic markers from adipose tissue (leptin, ghrelin, adiponectin).

We also aim to determine whether the hormonal response induced by orosensory stimulation by lipids is modified:

* in patients with type 2 diabetes
* in obese non-diabetic patients We expect to show an increase in biological markers biological, and more particularly in certain digestive hormones such as Pancreatic polypeptide, GIP, GLP-1…after stimulation of the lingual lipid receptor, CD36. We will also determine whether or not this response is modified in patients with type 2 diabetes and in obese non-diabetic patients.

We also wish to measure the subjects' gustatory detection threshold for a fatty acid (linoleic acid), and to determine whether there is a relationship between the orosensory perception threshold for linoleic acid and the physiological status of the subjects. In order to achieve this, the thresholds for healthy subjects will be compared with thresholds for obese and diabetic subjects. Expected results: the threshold of detection for linoleic acid in healthy subjects will be lower than that in obese or diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* Healthy volunteers:
* Men > 18 years
* 19 <BMI < 25 kg.m-2
* Fasting triglyceridemia < 1.50 g/l
* Fasting glycemia < 1.10 g/l
* Without regular medical treatment
* Patients with type-2 diabetes:
* Men >18 years
* type 2 diabetes (fasting glycemia > 7 mmol/l at the diagnosis) treated with diet or diet + oral antidiabetics (metformin, and/or insulinsecretion agents [hypoglycemic sulphonamides, or glinides] and/or glitazones and/or acarbose)
* Stable oral antidiabetic treatment for 3 months
* Obese non-diabetic patients:
* Men > 18 years
* BMI 30 kg.m-2
* Fasting glycemia < 1.10 g/l
* HbA1c < 6.0%
* Absence of treatment with hypoglycemic agents (including benfluorex)
* Absence of medical treatment for obesity
* Absence of a history of surgery for obesity (band, by-pass) or gastric stimulator (type Tantalus)

Exclusion Criteria:

* Persons not covered by the national health insurance
* Smokers, or smoking cessation within the 3 months preceding inclusion
* Persons with eating disorders:
* Severe digestive disease (enteropathy with absorption disorders, inflammatory digestive disease)
* Pancreatic insufficiency
* History of pancreas surgery
* Type 1 diabetes
* Renal insufficiency
* Hepatic insufficiency
* Treatment with proton pump inhibitors, insulin, GLP-1 analogues, DPP-4 inhibitors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2012-03-30 (Actual); Study Completion 2012-03-30 (Actual)

PRIMARY OUTCOMES:
Plasma levels of biological markers of orosensorielle perception fatty acids | Change from baseline at 15 days

SECONDARY OUTCOMES:
Measure the detection threshold for linoleic acid | baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France

REFERENCES:
- [Result] Chevrot M, Passilly-Degrace P, Ancel D, Bernard A, Enderli G, Gomes M, Robin I, Issanchou S, Verges B, Nicklaus S, Besnard P. Obesity interferes with the orosensory detection of long-chain fatty acids in humans. Am J Clin Nutr. 2014 May;99(5):975-83. doi: 10.3945/ajcn.113.077198. Epub 2014 Feb 12. PMID 24522446
- [Derived] Besnard P, Christensen JE, Bernard A, Simoneau-Robin I, Collet X, Verges B, Burcelin R. Identification of an oral microbiota signature associated with an impaired orosensory perception of lipids in insulin-resistant patients. Acta Diabetol. 2020 Dec;57(12):1445-1451. doi: 10.1007/s00592-020-01567-9. Epub 2020 Jul 16. PMID 32676702